CLINICAL TRIAL: NCT02544503
Title: Customized Cortical Stimulation Therapy in the Rehabilitation of Stroke Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was suspended in 2020 due to COVID-19 safety measures. Follow up with those previously enrolled later resumed, but not all subjects returned due to the ongoing pandemic. The study closed after attempting to obtain as much data as possible.
Sponsor: Emory University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Cathrin Buetefisch, Professor, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB00081238; R01NS090677 (NIH)
Record Dates: First submitted 2015-09-07; First posted 2015-09-09 (Estimated); Results first posted 2022-08-23 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Stroke
Keywords: Subacute stroke; Chronic stroke
MeSH Terms: conditions — Stroke | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Stroke Patients (Experimental): Subjects will undergo single pulse transcranial magnetic stimulation (TMS), paired pulse transcranial stimulation (ppTMS), and low frequency repetitive transcranial magnetic stimulation (rTMS) at one month and six months post stroke.
  Interventions: Device: Single-pulse Transcranial Magnetic Stimulation (TMS); Device: Paired-pulse Transcranial Magnetic Stimulation (ppTMS); Device: Low-frequency Repetitive Transcranial Magnetic Stimulation (rTMS); Device: Sham Motor Cortex Stimulation
- Healthy Controls (Active Comparator): Subjects will undergo single pulse transcranial magnetic stimulation (TMS), paired pulse transcranial stimulation (ppTMS), and low frequency repetitive transcranial magnetic stimulation (rTMS) at one month and six months.
  Interventions: Device: Single-pulse Transcranial Magnetic Stimulation (TMS); Device: Paired-pulse Transcranial Magnetic Stimulation (ppTMS); Device: Low-frequency Repetitive Transcranial Magnetic Stimulation (rTMS); Device: Sham Motor Cortex Stimulation

INTERVENTIONS:
Device: Single-pulse Transcranial Magnetic Stimulation (TMS) — Single-pulse Transcranial Magnetic Stimulation (TMS) is a brief magnetic pulse that is applied through a coil to the section of the head that overlays the motor cortex of the brain. Subjects will be comfortably seated in a dental chair surrounded by a frame that carries a coil holder to assist with the application of TMS to the brain. Single-pulse transcranial magnetic stimulation (TMS) will be administered at study visits.
Device: Paired-pulse Transcranial Magnetic Stimulation (ppTMS) — Paired-pulse Transcranial Magnetic Stimulation (ppTMS) is two brief sequential magnetic pulses that are applied through a coil to the section of the head that overlays the motor cortex of the brain. Subjects will be comfortably seated in a dental chair surrounded by a frame that carries a coil holder to assist with the application of TMS to the brain. Paired-pulse transcranial magnetic stimulation (ppTMS) will be administered at study visits.
Device: Low-frequency Repetitive Transcranial Magnetic Stimulation (rTMS) — Low-frequency Repetitive Transcranial Magnetic Stimulation (rTMS) is a sequence of brief magnetic pulses that are applied at 0.1 Hz frequency at low intensity through an air-cooled coil to the section of the head that overlays the motor cortex of the brain. Subjects will be comfortably seated in a dental chair surrounded by a frame that carries a coil holder to assist with the application of TMS to the brain. Low-frequency repetitive transcranial magnetic stimulation (rTMS) will be administered at study visits.
Device: Sham Motor Cortex Stimulation — Sham motor cortex stimulation will be applied at study visits.

SUMMARY:
The purpose of this study is to identify and establish how the area of the brain that controls motor function (motor cortex) of the non-affected hemisphere after stroke might serve as a new target for therapeutic interventions to improve motor performance after stroke.

DETAILED DESCRIPTION:
It is well known that the motor area of one hemisphere of the brain (motor cortex) controls the movement of the opposite side of the body but the role of the motor cortex in the hemisphere spared by stroke (contralesional motor cortex) in motor performance during post stroke recovery is still unclear. It is also not clear whether the motor cortex of both hemispheres of the brain are involved, as movement becomes more complicated. Currently the role of the motor cortex on the same side of the body (referred to as ipsilateral motor cortex) in hand performance remains controversial. In most patients with stroke, only one side of the brain is affected by the stroke (affected hemisphere) resulting in weakness of half of the body opposite to the side of the stroke. Over the recent years, research has discovered that the side of the brain, that is spared by the stroke (non-affected hemisphere) may support recovery after stroke. However, there is also a question whether the non-affected hemisphere may interfere with the process of recovery. It is currently not known what factors influence the activity of non-affected hemisphere to either support or interfere with the recovery of stroke. A better understanding of those events is critical to development of optimal therapeutic strategies. For example, non-invasive stimulation of specific areas of the non-affected hemisphere may help to improve functional recovery following stroke. The objectives of this study are to define the factors that influence the activity in the non-affected hemisphere to either support or interfere with the recovery after stroke. The researchers will study the area of the brain that controls movements of the non-affected hemisphere as it relates to motor function post-stroke.

Transcranial magnetic stimulation (TMS) is a device that allows non-invasive stimulation of the brain. When the brain is stimulated repetitively at a very low rate and low intensity for about 15 minutes, the stimulated brain area becomes less active. This effect lasts 10 minutes and is called a "transient artificial lesion" as it mimics the effects of transiently interfering with the function of the stimulated brain area. The study includes experiments that first identify the extent of stroke and brain areas involved in a motor task using functional MRI of the brain and TMS. The researchers will then determine the functional role of the contralesional motor cortex by studying the effect of low frequency and high frequency repetitive transcranial magnetic stimulation (rTMS) of primary motor cortex (M1) on interhemispheric inhibition (IHI) (resting and active) and motor cortex excitability (short interval intracortical excitability and corticospinal excitability) and behavior. The researchers will thereby also identify rTMS protocols that enhance motor performance in stroke patients.

In this study the researchers will conduct experiments using repetitive TMS to downregulate the activity of the motor area and measures its effect on activity of motor cortex of both hemispheres. In addition to enrolling participants who have had a stroke, the researchers will enroll healthy participants as this collected data will provide normative values for task related changes in M1s and their interactions - a prerequisite to studying abnormalities in stroke patients during motor recovery. The measurements and interventions will occur at two time points in all participants with stroke (1 and 6 months post-stroke). The data will be compared to the results of healthy age matched controls, assessed at a single time point.

ELIGIBILITY:
Inclusion Criteria for all Participants

* The ability to provide informed consent
* Ages 40 to 80 years old
* Male or female

Additional Inclusion Criteria for Stroke Patients:

* One cerebral ischemic infarction less than 1 month affecting the primary motor output system of the hand at a cortical (M1) level as defined by magnetic resonance imaging (MRI) of the brain
* Paresis of the hand for more than 3 days after their cerebral infarction

Additional Inclusion Criteria for Healthy Subjects:

* Normal MRI of the brain
* Normal neuropsychological testing
* Normal neurological examination

Exclusion Criteria for Stroke Patients:

* Neurological disorders other than stroke
* Aphasia that prevents following instructions or inability to communicate effectively with the study team
* Dementia
* Moderate or severe depression
* Contraindication to transcranial magnetic stimulation (TMS) and/or MRI
* Use of central nervous system (CNS) active drugs that block plasticity

Exclusion Criteria for Healthy Subjects:

* Neurological Disease
* Psychiatric Disease
* Use of CNS active drugs
* Contraindication to transcranial magnetic stimulation (TMS) and/or MRI

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-11-05 (Actual); Primary Completion 2021-02-04 (Actual); Study Completion 2021-02-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cathrin Buetefisch, MD, PhD, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Center for Rehabilitation Medicine, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Emory University School of Medicine, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Revill KP, Rizor E, Haut MW, Grafton ST, Buetefisch CM. Mean Motor Disconnectivity Predicts Hand Function Impairment After Stroke: Beyond Motor Cortex Output. Stroke. 2026 Jan 7:10.1161/STROKEAHA.125.052559. doi: 10.1161/STROKEAHA.125.052559. Online ahead of print. PMID 41498148
- [Derived] Wischnewski M, Edwards L, Revill KP, Drake D, Hobbs G, Buetefisch CM. Intensity-Dependent Effects of Low-Frequency Subthreshold rTMS on Primary Motor Cortex Excitability and Interhemispheric Inhibition in Elderly Participants: A Randomized Trial. Neurorehabil Neural Repair. 2025 Jan;39(1):58-73. doi: 10.1177/15459683241292615. Epub 2024 Oct 27. PMID 39462433
- [Derived] Buetefisch CM, Haut MW, Revill KP, Shaeffer S, Edwards L, Barany DA, Belagaje SR, Nahab F, Shenvi N, Easley K. Stroke Lesion Volume and Injury to Motor Cortex Output Determines Extent of Contralesional Motor Cortex Reorganization. Neurorehabil Neural Repair. 2023 Feb-Mar;37(2-3):119-130. doi: 10.1177/15459683231152816. Epub 2023 Feb 14. PMID 36786394

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at Emory University in Atlanta, Georgia, USA. Participant enrollment began in July 2015 and all follow-up assessments were completed by February 4, 2021.
Pre-assignment Details: Individuals provided consent to participate and were enrolled into study arms based on their health status (prior stroke or health control). After enrolling, 24 individuals with stroke and 3 healthy controls did not meet eligibility criteria and did not participate in any study assessments. Participants with stroke were assessed one and six months after their stroke, while healthy controls participated in a single assessment.
Groups:
- Stroke Patients: Participants with stroke underwent assessment of their upper extremity and hand motor function, MRI of their brain, single pulse transcranial magnetic stimulation (TMS), paired pulse transcranial stimulation (ppTMS), and low frequency repetitive transcranial magnetic stimulation (rTMS) at one month and six months post stroke.
- Healthy Controls: Healthy control participants underwent MRI, single pulse transcranial magnetic stimulation (TMS), paired pulse transcranial stimulation (ppTMS), and low frequency repetitive transcranial magnetic stimulation (rTMS).
Period: Overall Study
Arm/Group | Stroke Patients | Healthy Controls
Started | 66 | 34
Completed First Study Assessment (For stroke patients, the first study visit occurred one month after their stroke.) | 42 | 31
Stroke Patients Who Completed the 6 Month Post-stroke Assessment | 32 | 0 (Healthy control participants were not assessed at the 6 month time point.)
Completed | 32 | 31
Not Completed | 34 | 3
Not completed — Screen fail; these participants did not take part in the 1 month assessment | 24 | 3
Not completed — Lost to Follow-up | 9 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: The baseline analysis presented here includes participants who met eligibility criteria.
Groups:
- Total: Total of all reporting groups
Arm/Group | Stroke Patients | Healthy Controls | Total
Number analyzed (Participants) | 42 | 31 | 73
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.83 (9.43) | 61.68 (8.65) | 60.94 (9.21)
Age, Customized [Count of Participants; unit: Participants]
  Age, categorical: Less than 40 | 0 | 0 | 0
  Age, categorical: 40 - 80 | 42 | 31 | 73
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 17 | 40
  Male | 19 | 14 | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 24 | 8 | 32
  White | 14 | 4 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 19 | 21
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 42 | 31 | 73

OUTCOME MEASURES:

1. Primary Outcome: Motor Function Assessed by the Jebsen Test
Description: The Jebsen Test assesses weighted and non-weighted hand function among participants who have had a stroke. Subjects are assessed through writing, turning over 3 by 5 inch cards, picking up small common objects, simulated feeding, stacking checkers, picking up large objects, and picking up large heavy objects. Patients are required to perform all of the subtests with both the right and left hands. Time to complete each task is recorded and normalized to healthy age and sex matched control subjects. The score ranges from 0 to 1 with 0 being normal.
Time Frame: 1 month post-stroke (subacute stroke), 6 months post-stroke (chronic stroke)
Population: This analysis includes participants who completed this assessment at the indicated study visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stroke Patients
Number analyzed (Participants) | 32
score on a scale
  More affected hand - subacute stroke | 0.49 (0.32)
  Less affected hand - subacute stroke | 0.14 (0.10)
  More affected hand - chronic stroke: number analyzed (Participants) | 28
  More affected hand - chronic stroke | 0.35 (0.31)
  Less affected hand - chronic stroke: number analyzed (Participants) | 28
  Less affected hand - chronic stroke | 0.11 (0.09)

2. Primary Outcome: Mean Motor Evoked Potential (MEP) Amplitudes Assessed by Stimulus Response Curve (SRC) of the Contralesional M1
Description: Change in mean motor evoked potential (MEP) amplitudes at each stimulus intensity will be calculated. The sum of these means is calculated as the area under the curve.
Time Frame: 1 month post-stroke (subacute stroke) or single study visit for healthy controls, 6 months post-stroke (chronic stroke)
Population: This analysis includes participants completing the assessment at the indicated time point.
Measure: Mean (Standard Deviation); unit: mV
Arm/Group | Stroke Patients | Healthy Controls
Number analyzed (Participants) | 35 | 12
mV
  Subacute stroke or single visit for healthy controls | 0.67 (0.75) | 0.63 (0.85)
  Chronic stroke: number analyzed (Participants) | 19 | 0
  Chronic stroke | 0.39 (0.63) |

3. Primary Outcome: Presence of MEP in Response to TMS of the Ipsilesional M1
Description: The presence of motor evoked potential (MEP) in response to maximum TMS applied to ipsilesional M1 was determined in participants with stroke.
Time Frame: 1 month post-stroke (subacute stroke), 6 months post-stroke (chronic stroke)
Population: This analysis includes participants who completed the assessment at the indicated time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Stroke Patients
Number analyzed (Participants) | 35
Participants
  Subacute stroke: Not Present | 11
  Subacute stroke: Present | 24
  Chronic stroke: number analyzed (Participants) | 25
  Chronic stroke: Not Present | 3
  Chronic stroke: Present | 22

4. Primary Outcome: Lesion Volume
Description: Normalized stroke lesion volume was determined at the one-month time point using structural MRI of the brain.
Time Frame: 1 month post-stroke (subacute stroke)
Population: This analysis includes participants with stroke who completed this assessment.
Measure: Mean (Standard Deviation); unit: cubic mm
Arm/Group | Stroke Patients
Number analyzed (Participants) | 35
cubic mm | 19745 (32285)

5. Primary Outcome: Corticospinal Tract (CST) Lesion
Description: Corticospinal tract (CST) lesion load will be determined at the one-month time point using structural MRI of the brain. The lesion size is expressed as percentage of the entire CST.
Time Frame: 1 month post-stroke (subacute stroke)
Population: This analysis includes participants with stroke who completed this assessment.
Measure: Mean (Standard Deviation); unit: percent of CST
Arm/Group | Stroke Patients
Number analyzed (Participants) | 35
percent of CST | 5.7 (6.77)

6. Secondary Outcome: Motor Function Assessed by Time to Complete the Wolf Motor Function Test (WMFT)
Description: Upper extremity motor ability among participants who had a stroke was evaluated with the Wolf Motor Function Test (WMFT). The test consists of 17 items (6 joint-segment movements, 9 integrative functional movements and 2 strength items). The items are rated on a 6-point functional ability scale (FAS) where 0 is "no attempt is made to use the more affected arm and 5 is a normal appearance of movement execution. The time taken to complete each task will be recorded up to 120 seconds. The mean time to complete all tasks will be used to evaluate motor ability.
Time Frame: 1 month post-stroke (subacute stroke), 6 months post-stroke (chronic stroke)
Population: This analysis includes participants who completed this assessment at the indicated study visit.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Stroke Patients
Number analyzed (Participants) | 39
seconds
  Less affected side - subacute stroke | 7.11 (9.49)
  More affected side - subacute stroke | 36.82 (7.55)
  Less affected side - chronic stroke: number analyzed (Participants) | 26
  Less affected side - chronic stroke | 3.42 (4.86)
  More affected side - chronic stroke: number analyzed (Participants) | 26
  More affected side - chronic stroke | 18.44 (4.81)

7. Secondary Outcome: Motor Function Assessed by Grip Strength During the Wolf Motor Function Test (WMFT)
Description: During the grip strength assessment of the WMFT, participants grip a dynamometer with as much strength as possible. There are three trials of gripping with a minute rest interval between trials. The mean kilograms of strength exerted during the three trials is calculated.
Time Frame: 1 month post-stroke (subacute stroke), 6 months post-stroke (chronic stroke)
Population: This analysis includes participants completing the assessment at the indicated time point.
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Stroke Patients
Number analyzed (Participants) | 39
kilograms
  Less affected side - subacute stroke | 28.95 (10.88)
  More affected side - subacute stroke | 15.25 (15.70)
  Less affected side - chronic stroke: number analyzed (Participants) | 26
  Less affected side - chronic stroke | 29.94 (8.06)
  More affected side - chronic stroke: number analyzed (Participants) | 26
  More affected side - chronic stroke | 17.03 (12.68)

8. Secondary Outcome: Use of Paretic Arm Assessed by the Motor Activity Log (MAL)
Description: In stroke patients, the everyday use of the paretic (the more affected) arm will be measured using the Motor Activity Log (MAL). The MAL is a subjective measure of semi- structured interview to examine a) how much and b) how well the subject uses their more-affected arm outside of the laboratory setting. Total scores range from 0 (no use of the more-affected arm) to 5 (use is as good as before stroke).
Time Frame: 1 month post-stroke (subacute stroke), 6 months post-stroke (chronic stroke)
Population: This analysis includes participants with stroke who completed the assessment during the indicated study visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stroke Patients
Number analyzed (Participants) | 35
score on a scale
  Amount of use, subacute stroke | 2.044 (1.654)
  Quality of movement, subacute stroke | 1.939 (1.593)
  Amount of use, chronic stroke: number analyzed (Participants) | 30
  Amount of use, chronic stroke | 3.266 (1.625)
  Quality of movement, chronic stroke: number analyzed (Participants) | 30
  Quality of movement, chronic stroke | 3.275 (1.597)

9. Secondary Outcome: CST Subpathway Originating in M1 Lesion Load
Description: CST sub M1 lesion volume will be determined at the one- month time point using structural MRI of the brain. The lesion load is expressed as percentage of the entire CST.
Time Frame: 1 month post-stroke (subacute stroke)
Population: This analysis includes participants with stroke who completed this assessment.
Measure: Mean (Standard Deviation); unit: percentage of the entire CST
Arm/Group | Stroke Patients
Number analyzed (Participants) | 35
percentage of the entire CST | 5.07 (6.48)

10. Secondary Outcome: Primary Motor Cortex (M1) Activity, Assessed by Functional Magnetic Resonance Imaging (fMRI)
Description: Functional Magnetic Resonance Imaging (fMRI) will be used to determine hand movement related activity in the motor cortex of the brain in all subjects. Blood oxygenation level dependent (BOLD) response during execution of the motor task will be compared to rest. The subacute stroke and chronic stroke time points are compared to single study visit of healthy controls.
Time Frame: 1 month post-stroke (subacute stroke) or single study visit for healthy controls, 6 months post-stroke (chronic stroke)
Population: This analysis includes participants completing the assessment at the indicated time point.
Measure: Mean (Standard Deviation); unit: Percent signal change
Arm/Group | Stroke Patients | Healthy Controls
Number analyzed (Participants) | 19 | 31
Percent signal change
  Ipsilesional - subacute stroke: number analyzed (Participants) | 19 | 0
  Ipsilesional - subacute stroke | 1.33 (1.10) |
  Contralesional - subacute stroke: number analyzed (Participants) | 19 | 0
  Contralesional - subacute stroke | 0.14 (0.41) |
  Contralateral Left - single visit for healthy controls: number analyzed (Participants) | 0 | 31
  Contralateral Left - single visit for healthy controls |  | 1.59 (0.75)
  Contralateral Right - single visit for healthy controls: number analyzed (Participants) | 0 | 31
  Contralateral Right - single visit for healthy controls |  | 1.59 (0.82)
  Ipsilateral Left - single visit for healthy controls: number analyzed (Participants) | 0 | 31
  Ipsilateral Left - single visit for healthy controls |  | 0.27 (0.55)
  Ipsilateral Right - single visit for healthy controls: number analyzed (Participants) | 0 | 31
  Ipsilateral Right - single visit for healthy controls |  | 0.17 (0.36)
  Ipsilesional - chronic stroke: number analyzed (Participants) | 12 | 0
  Ipsilesional - chronic stroke | 0.68 (0.52) |
  Contralesional - chronic stroke: number analyzed (Participants) | 12 | 0
  Contralesional - chronic stroke | 0.03 (0.27) |

11. Secondary Outcome: Short Interval Cortical Inhibition (SICI) Measured by Repeated Transcranial Magnetic Stimulation (rTMS)
Description: SICI in the contralesional M1 will be measured using paired pulse TMS at an interstimulus interval (ISI) of 2 milliseconds (ms). Cortical stimulation intensity was delivered at 60% and 80% of the motor threshold (MT). SICI is expressed as the ratio between the mean MEP amplitude in response to a single TMS and the mean MEP amplitude in response to a paired pulse TMS. A ratio of 1 means no inhibition, a ratio smaller than 1 means inhibition, and a ratio greater than 1 means facilitation.
Time Frame: 1 month post-stroke (subacute stroke) or single study visit for healthy controls, 6 months post-stroke (chronic stroke)
Population: This analysis includes participants completing the assessment at the indicated study visit.
Measure: Mean (Standard Deviation); unit: ratio of MEP amplitude with TMS pulses
Arm/Group | Stroke Patients | Healthy Controls
Number analyzed (Participants) | 31 | 12
ratio of MEP amplitude with TMS pulses
  Sham Cortex Stimulation 60% MT, Pre - subacute stroke, or healthy control visit | 0.92 (0.70) | 1.00 (0.56)
  Sham Cortex Stimulation 60% MT, Post - subacute stroke, or healthy control visit | 0.76 (0.57) | 0.73 (0.32)
  Sham Cortex Stimulation 80% MT, Pre - subacute stroke, or healthy control visit | 0.93 (0.53) | 0.73 (0.68)
  Sham Cortex Stimulation 80% MT, Post - subacute stroke, or healthy control visit | 0.79 (0.36) | 0.56 (0.35)
  rTMS Cortex Stimulation 60% MT, Pre - subacute stroke, or healthy control visit | 0.84 (0.65) | 0.98 (0.64)
  rTMS Cortex Stimulation 60% MT, Post - subacute stroke, or healthy control visit | 0.92 (0.52) | 0.99 (0.42)
  rTMS Cortex Stimulation (CS) 80% MT, Pre - subacute stroke, or healthy control visit | 1.00 (0.55) | 0.88 (0.82)
  rTMS Cortex Stimulation (CS) 80%, Post - subacute stroke, or healthy control visit | 0.84 (0.58) | 0.77 (0.52)
  Sham Cortex Stimulation 60% MT, Pre - chronic stroke: number analyzed (Participants) | 19 | 0
  Sham Cortex Stimulation 60% MT, Pre - chronic stroke | 0.95 (0.68) |
  Sham Cortex Stimulation 60% MT, Post - chronic stroke: number analyzed (Participants) | 19 | 0
  Sham Cortex Stimulation 60% MT, Post - chronic stroke | 0.89 (0.43) |
  Sham Cortex Stimulation 80% MT, Pre - chronic stroke: number analyzed (Participants) | 19 | 0
  Sham Cortex Stimulation 80% MT, Pre - chronic stroke | 1.12 (0.69) |
  Sham Cortex Stimulation 80% MT, Post - chronic stroke: number analyzed (Participants) | 19 | 0
  Sham Cortex Stimulation 80% MT, Post - chronic stroke | 0.83 (0.54) |
  rTMS Cortex Stimulation 60% MT, Pre - chronic stroke: number analyzed (Participants) | 19 | 0
  rTMS Cortex Stimulation 60% MT, Pre - chronic stroke | 0.92 (0.71) |
  rTMS Cortex Stimulation 60% MT, Post - chronic stroke: number analyzed (Participants) | 19 | 0
  rTMS Cortex Stimulation 60% MT, Post - chronic stroke | 0.89 (0.99) |
  rTMS Cortex Stimulation (CS) 80% MT, Pre - chronic stroke: number analyzed (Participants) | 19 | 0
  rTMS Cortex Stimulation (CS) 80% MT, Pre - chronic stroke | 0.99 (0.46) |
  rTMS Cortex Stimulation (CS) 80%, Post - chronic stroke: number analyzed (Participants) | 19 | 0
  rTMS Cortex Stimulation (CS) 80%, Post - chronic stroke | 1.09 (0.46) |

12. Secondary Outcome: Peak Velocity During Wrist Extension Movement
Description: Stroke patients are asked to rapidly execute 7 ballistic wrist extension movements following an auditory cue. A 2-dimensional gyrometer is mounted on the dorsum of the hand to measure wrist extension movements. Electromyography (EMG) activity will be recorded on the extensor carpi ulnaris (ECU) muscle, a muscle that supports wrist extension movements.
Time Frame: 1 month post-stroke (subacute stroke), 6 months post-stroke (chronic stroke)
Population: This analysis includes participants with stroke who completed this assessment at the indicated study visit.
Measure: Mean (Standard Deviation); unit: radian per second (rad/sec)
Arm/Group | Stroke Patients
Number analyzed (Participants) | 35
radian per second (rad/sec)
  Less affected side - subacute stroke - rTMS pre | 700.54 (248.34)
  Less affected side - subacute stroke - rTMS post | 686.24 (305.79)
  Less affected side - subacute stroke - sham pre | 641.29 (280.48)
  Less affected side - subacute stroke - sham post | 628.23 (264.45)
  More affected side - subacute stroke - rTMS pre | 389.08 (313.69)
  More affected side - subacute stroke - rTMS post | 373.75 (294.01)
  More affected side - subacute stroke - sham pre | 413.10 (317.41)
  More affected side - subacute stroke - sham post | 398.41 (301.56)
  Less affected side - chronic stroke - rTMS pre: number analyzed (Participants) | 24
  Less affected side - chronic stroke - rTMS pre | 659.25 (266.67)
  Less affected side - chronic stroke - rTMS post: number analyzed (Participants) | 24
  Less affected side - chronic stroke - rTMS post | 630.80 (276.10)
  Less affected side - chronic stroke - sham pre: number analyzed (Participants) | 24
  Less affected side - chronic stroke - sham pre | 670.80 (269.49)
  Less affected side - chronic stroke - sham post: number analyzed (Participants) | 24
  Less affected side - chronic stroke - sham post | 653.85 (257.50)
  More affected side - chronic stroke - rTMS pre: number analyzed (Participants) | 24
  More affected side - chronic stroke - rTMS pre | 430.58 (286.32)
  More affected side - chronic stroke - rTMS post: number analyzed (Participants) | 24
  More affected side - chronic stroke - rTMS post | 415.61 (290.76)
  More affected side - chronic stroke - sham pre: number analyzed (Participants) | 24
  More affected side - chronic stroke - sham pre | 444.48 (288.84)
  More affected side - chronic stroke - sham post: number analyzed (Participants) | 24
  More affected side - chronic stroke - sham post | 440.02 (294.17)

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected beginning at the first study visit and continued through the final assessment, up to one year.
Arm/Group | Stroke Patients | Healthy Controls
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/31
Other Adverse Events (participants affected / at risk) | 14/42 | 1/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stroke Patients (N=42) | Healthy Controls (N=31)
Headache (General disorders) | 5 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 8 | 0
Panic attack in MR (Psychiatric disorders) | 1 | 0
Soreness in the wrist (Musculoskeletal and connective tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-10-01): https://cdn.clinicaltrials.gov/large-docs/03/NCT02544503/Prot_SAP_000.pdf
  • Informed Consent Form (2019-10-01): https://cdn.clinicaltrials.gov/large-docs/03/NCT02544503/ICF_001.pdf